CLINICAL TRIAL: NCT04557800
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Of DNL151 in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL151 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-C-0001; 2017-003730-82 (EudraCT Number)
Record Dates: First submitted 2020-09-10; First posted 2020-09-22 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — DNL151

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DNL151 (Experimental): Part A: Single-ascending dose cohorts; Part B: Multiple-ascending dose cohorts (10 days); Part C: Single-dose cohort; Part D: Additional multiple-dose cohort (28 days); Part E Multiple-ascending dose cohorts (14 days)
  Interventions: Drug: DNL151
- Placebo (Placebo Comparator): Part A: Single-ascending dose cohorts; Part B: Multiple-ascending dose cohorts (10 days); Part C: Single-dose cohort; Part D: Additional multiple-dose cohort (28 days); Part E Multiple-ascending dose cohorts (14 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNL151 — oral dose(s)
  Arms: DNL151
Drug: Placebo — oral dose(s)
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose (SAD), multiple ascending dose (MAD), and 28-day safety study of orally administered DNL151 in healthy volunteers.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under Section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by Sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index 18.5 to 35.0 kg/m², inclusive, and body weight of at least 50.0 kg at screening
* In good health, determined by no clinically significant findings from medical history, physical examination, and vital sign measurements
* Women of non-childbearing potential and men using contraceptive measures

Key Exclusion Criteria:

* History of clinically significant hematological, renal, pancreatic, gastrointestinal, hepatic, cardiovascular, metabolic, endocrine, immunological, allergic disease, or other major disorders
* History of asthma, chronic obstructive pulmonary disease, or emphysema
* Clinically significant neurologic disorder
* History of stomach or intestinal surgery or resection
* History of malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs), and discontinuations due to TEAEs | Up to 42 days
PK parameter: Maximum observed concentration (Cmax) of DNL151 in plasma | Up to 42 days
PK parameter: Time to maximum observed concentration (Tmax) of DNL151 in plasma | Up to 42 days
PK parameter: The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of DNL151 in plasma (single dosing only) | Up to 42 days
PK parameter: Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC[0-last]) of DNL151 in plasma | Up to 42 days
PK parameter: The area under the concentration-time curve over a dosing interval (AUC0-τ) of DNL151 in plasma (multiple dosing only) | Up to 42 days
PK parameter: Apparent terminal elimination half-life (t1/2) of DNL151 in plasma | Up to 42 days

SECONDARY OUTCOMES:
Concentration of DNL151 in cerebrospinal fluid (CSF) (following selected single and multiple doses) | Up to 13 days
The pharmacodynamics of DNL151 in whole blood as measured by the percent change from baseline in pS935 | Up to 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Andres Cruz-Herranz, Study Director — Denali Therapeutics Inc.
Locations (2):
- Netherlands (2):
  - Centre for Human Drug Research, Leiden, South Holland
  - PRA Health Sciences, Van Swietenlaan, Groningen

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102